CLINICAL TRIAL: NCT03081312
Title: A Study of Family Caregivers' Needs, Burden of Care and Quality of Life Over the Course of a Cancer Illness
Acronym: FCG-NBC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, Rathi Mahendran, Principal Investigator, National University of Singapore
Other Study IDs: 2017/00029
Record Dates: First submitted 2017-03-07; First posted 2017-03-16 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-01

CONDITIONS: Family Caregivers; Cancer; Health Related Quality of Life
Keywords: Family Cancer Caregivers,; Needs; Burden of Care; Quality of Life
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This research will determine (a) the unmet needs of family caregivers of adult cancer patients and (b) determine the impact on stress, care burden and quality of life.

A cross-sectional questionnaire methodology will be used to answer the research questions. 510 family caregivers at different stages of patients' cancer journey will be recruited. The study duration is expected to take two years. Research findings will address the knowledge gap of caregivers' needs and stress, burden and quality of life and support plans to help caregivers.

DETAILED DESCRIPTION:
The literature suggests that caregivers have unique psychological, emotional and lifestyle needs but there is a paucity of such information of caregivers in Singapore. As this study is exploratory, no a priori hylothesis has been made. The theoretical framework guiding this research is Fulfillment Theory in which the existence and perception of needs and need fulfillment are hypothesized to be antecedents to the experience of satisfaction about care.

A cross-sectional questionnaire methodology will be used to answer the research questions. Caregivers in this study are defined as: a family member who lends physical, emotional or other support to someone at any time during the cancer journey. A power calculation was not done, instead the sample size of 510 was based on what may be practically achievable and feasible for the duration of the short-term quantitative study. Descriptive statistics will be used to characterize the distribution of socio-demographic characteristics and caregiver-related information. Regression analysis will be used to evaluate difference in overall and domain specific needs across selected characteristics. Problems identified by caregivers will be dichotomized as present or absent and chi-square tests will be used to evaluate associations with selected characteristics.

ELIGIBILITY:
Inclusion Criteria:

an adult providing care for a familyt member with cancer aged between 21 and 90 years and willing to participate in the study

Exclusion Criteria:

caregiving adults who are not family members and not willing to particfipate in the study

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Family cancer caregiver - defined as a family member who lends physical, emotional or other support to someone at any time during cancer treatment.
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-02-28 (Estimated)

PRIMARY OUTCOMES:
Needs of family cancer caregivers | One year
  Needs Assessment of Family Caregivers-Cancer (NAFC-C) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, MMed(Psych), Principal Investigator — Department of Psychological medicine, NUS
Locations (1):
- Department of Psychological Medicine, NUS, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No